CLINICAL TRIAL: NCT05692362
Title: Measure Airway Compliance by Endobronchial Optical Coherence Tomography
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Xu Hang, Dierctor of Intervetional Pulmonary Center, The First Affiliated Hospital of Guangzhou Medical University
Other Study IDs: GYFYY20221108
Record Dates: First submitted 2023-01-04; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Tomography, Optical Coherence; Bronchoscopy; Respiratory Disease; Airway Remodeling
Keywords: EB-OCT; Airway Compliance; Airway Remodeling
MeSH Terms: conditions — Respiration Disorders; Airway Remodeling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Airway Biopsy for IHC
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- Healthy People: People with solitary pulmonary nodule， without any other pulmonary diseases.
- Chronic Airway Diease People: People with COPD or Asthma
- Pulmonary fibrosis people: People were diagnosised pulmonary fibrosis by chest Computer Tomography, and restrictive ventilatory impairment by pulmonary function test.

SUMMARY:
Optical Coherence Tomography （OCT）is a novel, non-invasive, high resolution special optical imaging techniques. In airway, Measure airway area and airway wall thickness is the most usage of Endobronchial Optical Coherence Tomography (EB-OCT）. Recently, the new protocol of EB-OCT is used to measure airway compliance, We will establish a new methodology of EB-OCT for measuring airway compliance, which will provide a new means to study respiratory diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Regardless of gender, age 18-70 years old;
2. Patients with clinical diagnosis of pulmonary nodules, COPD, asthma or restrictive pulmonary diseases;
3. Can tolerate bronchoscopy patients;
4. Sign the informed consent form.

Exclusion Criteria:

1. Suffering from any of the following respiratory diseases: bronchiectasis, etc;
2. Have malignant tumors that are not completely remission or cured;
3. The patient's systemic infection is not controlled;
4. Recent use of immunosuppressants, recent use of anticoagulants (such as warfarin or aspirin within 2 weeks of drugs that affect blood clotting function);
5. Serious other systemic diseases: myocardial infarction, unstable angina, cirrhosis, acute glomerulonephritis, etc.;
6. Those who are positive for syphilis, HIV, HBV, and HCV antibodies;
7. Patients with coagulation dysfunction diseases, such as hemophilia, giant platelet syndrome, platelet weakness, etc.;
8. Severe renal impairment, serum creatinine > 1.5 times the upper limit of normal value;
9. Liver disease or liver function impairment: ALT, AST, total bilirubin > 2 times the upper limit of normal value;
10. Those with a history of mental illness or suicide, a history of epilepsy or other central nervous system diseases;
11. 12-lead ECG showing severe arrhythmias (such as ventricular tachycardia, frequent supraventricular tachycardia, atrial fibrillation, atrial flutter, etc.) or conduction abnormalities of the heart of grade II and above;
12. Those who are allergic to catheters and related materials required for experiments;
13. Subjects who have received any other clinical studies within 3 months prior to enrollment;
14. Those who have poor compliance and difficulty in completing the study;
15. Any condition that the clinician believes may increase the risk to the patient or interfere with the clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy People and People with COPD or asthma 、 restrictive pulmonary diseases.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Airway Compliance of different airway generation | 2023/01/01-2024/12/31
  Airway compliance is the property of the airway lumen area to change as pressure changes. This is caused by airway structure, the small airway without cartilage compared with medium and large airways, so the compliance would be different.
  But the methods of measuring airway compliance is difficult, In this research, we will use OCT to measure airway area (mm2), and record the airway pressure(cmH2O), The ratio of area change to pressure change is the compliance, we will measure and compare the compliance of different airway generation.

SECONDARY OUTCOMES:
Airway Compliance of different people | 2023/01/01-2024/12/31
  Airway compliance is the property of the airway lumen area to change as pressure changes. This is caused by airway structure, the airway of COPD, asthma or pulmonary fibrosis compared to healthy people are different, so the compliance would be different.
  But the methods of measuring airway compliance is difficult, In this research, we will use OCT to measure airway area (mm2), and record the airway pressure(cmH2O), The ratio of area change to pressure change is the compliance, we will measure and compare the compliance of different people.

CONTACTS AND LOCATIONS:
Locations (1):
- Hang Xu, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No